CLINICAL TRIAL: NCT05008471
Title: Application of Whole-course Standardized Nutrition Management During Peri-radiotherapy in Patients With Nasopharyngeal Carcinoma After Radiotherapy: a Multicenter Randomized Controlled Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Principal Investigator, Sun Yat-sen University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020-FXY-487
Record Dates: First submitted 2021-08-03; First posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Nasopharyngeal Carcinoma; Radiation Therapy Induced Change; Nutrition Disorders
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The recommended target energy for NPC radiotherapy patients is 25-30kcal/(kg·d), in addition，the intervention group begins with an additional 50% daily energy increase during the peri-radiotherapy.
  Interventions: Dietary Supplement: Formula nutrition
- Conventional group (No Intervention): Unlike the intervention group,conventional group should be treated according to the consensus of experts on standardized nutrition management.

INTERVENTIONS:
Dietary Supplement: Formula nutrition — The target energy of radiotherapy patients is recommended to be 25-30kcal/(kg·d), and the target energy of the intervention group should be increased by an additional 50% daily from the beginning of radiotherapy. Specifically, under the condition of ensuring the daily target energy 14kcal/(kg·d), formula nutrition should be added daily.
  Arms: Intervention group

SUMMARY:
This study will present an advanced equipment of tumor nutrition diagnosis and assesment for nasopharyngeal cancer(NPC) radiotherapy patients in nutritional risk screening, evaluation, diagnosis and directing nutritional intervention, aiming to explore the advantages of the whole nutritional management in acute radiation reaction rate, completion rate of radiotherapy, nutritional status, and quality of life for NPC patients.

DETAILED DESCRIPTION:
In this study, nutrition intervention was performed in one group of nasopharyngeal carcinoma patients with no nutritional risk during the periperiod of radiotherapy , and the other group with no additional intervention when without nutritional risks, for evaluating the value of overall nutritional management in the periperiod radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nasopharyngeal carcinoma confirmed by histopathology
* Newly diagnosed patients without distant metastasis
* Age >18
* KPS ≥ 70
* Nasopharyngeal radiotherapy alone or concurrent chemoradiotherapy was planned to be received, andIMRT was used for radiotherapy
* The patient's blood counts，the lung, liver and renal functions were tolerant to radiotherapy/chemoradiotherapy（ WBC ≥ 4.0*109/L, NE ≥ 2.0*109/L, PLT 100*109/L and Hb≥ 10g/L. AST and ALT ≤ 2.5 *the upper limit（UL） ,TBIL≤1.2*the UL, CRE≤1.2* the UL, and ALP≤5* the UL）. And the ECG should be normal
* Good nutritional status,BMI:18~23Kg/ m2, PG-SGA ≤1,NRS 2002<3score
* No other previous neoplastic diseases, except for cured cervical carcinoma in situ skin basal carcinoma
* No serious gastrointestinal diseases (moderate and severe duodenal and gastric ulcer, ulcerative colitis, Crohn's disease, etc.)
* No AIDS and no diabetes
* Clear mind, no communication barriers, able to answer questions
* Voluntarily participate and sign the informed consent in person.

Exclusion Criteria:

* Patients with gastrointestinal dysfunction, intestinal obstruction, pyloric obstruction, Acute gastrointestinal bleeding
* Patients who are allergic to nutritional therapy or have severe allergic constitution
* Uncontrolled systemic diseases, such as severe liver disease (such as cirrhosis), kidney disease, respiratory diseases and so on.
* Women who are pregnant or breastfeeding or no contraception and women with positive pregnancy test before receiving treatment
* Special dietary requirements: such as no having a certain food or a vegetarian.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2022-04-26 (Estimated); Study Completion 2022-04-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute radiation reactions | 12 months
  This study mainly includes oral mucosa mucositis, salivary glands injury induced by radiotherapy, laryngoesophageal mucositis referring to The 2020 Expert Consensus on the Standardized Management of Radiation Oncology for nutrition-related radiation injury responses.

SECONDARY OUTCOMES:
Incidence of decline in nutritional status | 12 months
  analysis by the clinical nutrition detection analyzer
Incidence of decline in quality of life scores（QOL） | 12 months
  It is measured by a standard QOL table,including 12 questions.Each question is 5 points,so there are 60 points and 5 grades(51-60 points, 41-50 points, 31-40 points, 21-30 points,<20 points).A higher score is a better life.
Self-rating Anxiety screening Scale（GAD-7) | 12 months
  A GAD-7 table would estimate one's anxiety according to the emotion of the past two weeks,including 9 questions and 27 points totally.There are 4 grades of anxiety, a LOWER score means a normal mind state. Actually,0-4 points is/are no anxiety.5-9 points represent slight anxiety .10-14 are in moderate anxiety.15-27 are severe anxiety,respectively.
Self-rating Scale for Depression Screening (PHQ-9) | 12 months
  A PHQ-9 table is a simplified Scale for Depression Screening,it would estimate one's depression emotion according to the mind of the past two weeks,including 9 questions and 27 points totally.There are 4 grades of depression, a LOWER score is equal to a GOOD mind.Actually,0-4 points is/are no depression.5-9 are depressed but not obvious.10-14 are in obvious depression.15-27 are severe depression,respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Xia, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangdong, Guangzhou, China